CLINICAL TRIAL: NCT01694537
Title: The Effects of DLBS1033 on Haemostasis Parameters in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Dexa Medica Group (Industry)
Responsible Party: Principal Investigator, Nafrialdi, MD, PhD, SpPD, SpFK, Indonesia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DLBS1033
Record Dates: First submitted 2012-09-07; First posted 2012-09-27 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: lumbrokinase; fibrinolytic; plasmin-antiplasmin complex; euglobulin clot lysis time; platelet aggregation
MeSH Terms: interventions — DLBS 1033

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): The comparison drug is placebo, which is made with same size and shape with study drug. DLBS1033 and placebo is produced by PT Dexa Medica. Placebo will taken 3 times 1 tablet per day for 7 days. Wash out period before enter another arm is 7 days.
  Interventions: Drug: DLBS1033; Drug: placebo
- DLBS1033 (Experimental): The study drug is enteric coated DLBS1033, which contain 490 mg bioactive protein fraction. The drug will taken 3 times 490 mg per day for 7 days. Wash out period before enter another arm is 7 days.
  Interventions: Drug: DLBS1033; Drug: placebo

INTERVENTIONS:
Drug: DLBS1033 — The study drug is enteric coated DLBS1033, which contain 490 mg bioactive protein fraction.
Drug: placebo — Placebo is made with same size and shape with study drug.

SUMMARY:
DLBS1033 is bioactive protein fraction which extracted from Lumbricus rubellus earthworm. This earthworm comes from Pengalengan, West Java, Indonesia. DLBS1033 possesses 8 major proteins with molecular weight below 100 kDa, so its named as Lumbricus Low Molecular weight Proteins (LLP). This enzym can be transported to the bloodstream via intestinal epitel. Structure of DLBS1033 looks like lumbrokinase. Lumbrokinase is enzym that consist of 6 isoenzyme serine protease. As a drug that consists of serin protease enzym, suspected that the mechanism of action of DLBS1033 similar with lumbrokinase, especially as plasminogen activator in fibrinolytic system. In vitro study by Trisina et al showed that DLBS1033 has fibrinogenolytic activities on fibrinogen α, beta, and gamma chain, decreasing platelet aggregation and clotting time was prolonged. Until now, the mechanism of action and effects of DLBS1033 on human fibrinolytic and coagulation system still unknown. Therefore, the aim of this clinical trial is to evaluate the effects of DLBS1033 on human fibrinolytic and coagulation system on healthy subjects.

DETAILED DESCRIPTION:
Fibrinolysis is a process to lyse clot formed by thrombin. It starts with activating plasminogen to plasmin by the endogenous tissue plasminogen activator (tPA) and urokinase plasminogen activator (uPA). These activator are found in the endothelium, granulocytes and monocytes. Plasminogen activator inhibitor-1 (PAI-1) is the major inhibitor of tPA and uPA) and α2-antiplasmin is major inhibitor of plasmin. Plasmin wil degrade soluble fibrinogen and fibrin to produce fibrinogen degradation products and fibrin degradation products, respectively.

Lumbrokinase has been investigated in animal studies. Kim et al was conducting on rats by administered freeze-dried powder of Lumbricus rubellus earthworm orally. This study showed that earthworm powder is valuable for the prevention and/or treatment of thrombotic conditions. Similar conclusion also shown on study by Lee et al, which compared antithrombotic and fibrinolytic activities of lumbrokinase SPP-501 (extracted from Eisenia andrei earthworm) with urokinase and t-PA in a thrombosis model of rat vena. The results of this study were decreasing of thrombus weight, shortening of euglobulin lysis time (ELT), and reducing platelet aggregation of rat which given SPP-501.

Conclusion from several clinical trial similar with several studies on animal. From study which was conducted by Jin et al on 51 cerebral infarct subjects which were given 3 times 400 mg lumbrokinase (n = 31) or control (n = 20) for 28 days. In the treatment group, kaolin partial thromboplastin time (KPTT) was prolonged, t-PA activity and D-dimer level increase, and fibrinogen decreased significantly. It is concluded that mechanism of lumbrokinase as oral antithrombotic and fibrinolytic are by inhibition of coagulation intrinsic pathway and activate fibrinolytic pathway by increasing t-PA activity. Fibrinolytic activity was also concluded by Rey, who was conducted study on 28 diabetic foot ulcer subjects, which were given 3 times 500 mg lumbrokinase per day (n = 14) for 7 days, or placebo. On this study, in the treatment group mean of D-dimer was increased.

From many clinical trials, it is concluded that effects of lumbrokinase have seen after several days. It is different with intravenous fibrinolytic enzym, such as streptokinase and t-PA, which effects have seen soon after it was used. Therefore oral lumbrokinase could not replace the function of intravenous fibrinolytic enzym,that was used on acute thrombosis. Based on antithrombotic and fibrinolytic activity, lumbrokinase might used as secondary prevention after acute thrombosis, such as myocard infarct and stroke. Some researchers have started clinical trials about that hypothesis.

Pilot study by Kasim et al was used a lumbrokinase in 10 patient with stable angina pectoris. This study showed that 70% of total sample receiving lumbrokinase had a significant decrease in summed stress score of perfusion imaging and better perfusion in viable myocardium after 30 days of lumbrokinase treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-55 years old
* body mass index between 18-25 kg/square metres
* normal physical examination
* Patient still have the ability to undergo examinations and give written informed consent
* Plasmin-antiplasmin complex (PAP complex) level between 0-514 ng/ml
* Platelet aggregation (ADP 10 uM) > 49%

Exclusion Criteria:

* Patient with cardiovascular disease, hypertension, diabetes mellitus, and dyslipidemia
* Creatinin serum more than 1,5 x upper limit normal
* SGOT and SGPT more than 3 x upper limit normal
* Blood pressure ≥ 140/90 mmHg
* Fasting blood glucose > 126 mg/dL
* Alcohol patients
* Took any medications (including traditional medicine, supplement and vitamin) in 1 week before the study)
* Patient has bleeding history which unclear etiology
* Hemoglobin < 10 g/dL
* Thrombocyte count < 100.000/uL
* Heavy smoker (Bringman Index > 600)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
plasmin-antiplasmin complex (PAP complex) | one week
  changes in plasmin-antiplasmin complex

SECONDARY OUTCOMES:
euglobulin clot lysis time (ECLT) | one week
  changes in euglobulin clot lysis time
prothrombin time (PT) | one week
  changes in prothrombin time
fibrinogen | one week
  changes in fibrinogen
activated partial thromboplastin time (aPTT) | one week
  changes in activated partial thromboplastin time
platelet aggregation | one week
  changes in platelet aggregation

OTHER OUTCOMES:
serum creatinine | one week
  serum creatinine
serum glutamic oxaloacetic transaminase (SGOT) | one week
  changes in serum glutamic oxaloacetic transaminase
serum glutamic pyruvic transaminase (SGPT) | one week
  changes in serum glutamic pyruvic transminase

CONTACTS AND LOCATIONS:
Overall Officials: Nafrialdi, MD, PhD, SpPD, SpFK, Principal Investigator — Indonesia University
Locations (1):
- Indonesia University, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mihara H, Sumi H, Yoneta T, Mizumoto H, Ikeda R, Seiki M, Maruyama M. A novel fibrinolytic enzyme extracted from the earthworm, Lumbricus rubellus. Jpn J Physiol. 1991;41(3):461-72. doi: 10.2170/jjphysiol.41.461. PMID 1960890
- [Background] Kasim M, Kiat AA, Rohman MS, Hanifah Y, Kiat H. Improved myocardial perfusion in stable angina pectoris by oral lumbrokinase: a pilot study. J Altern Complement Med. 2009 May;15(5):539-44. doi: 10.1089/acm.2008.0506. PMID 19416019
- [Background] Yan XM, Kim CH, Lee CK, Shin JS, Cho IH, Sohn UD. Intestinal Absorption of Fibrinolytic and Proteolytic Lumbrokinase Extracted from Earthworm, Eisenia andrei. Korean J Physiol Pharmacol. 2010 Apr;14(2):71-5. doi: 10.4196/kjpp.2010.14.2.71. Epub 2010 Apr 30. PMID 20473377
- [Result] Lee CK, Shin JS, Kim BS, Cho IH, Kim YS, Lee EB. Antithrombotic effects by oral administration of novel proteinase fraction from earthworm Eisenia andrei on venous thrombosis model in rats. Arch Pharm Res. 2007 Apr;30(4):475-80. doi: 10.1007/BF02980222. PMID 17489364
- [Result] Kim YS, Pyo MK, Park KM, Hahn BS, Yang KY, Yun-Choi HS. Dose dependency of earthworm powder on antithrombotic and fibrinolytic effects. Arch Pharm Res. 1998 Aug;21(4):374-7. doi: 10.1007/BF02974629. PMID 9875462
- [Result] Schmaier AH, Thornburg CD, Pipe SW. Coagulation and Fibrinolysis. In: McPherson RA, Pincus MR, editor. Henry's Clinical Diagnosis and Management by Laboratory Methods. 21st ed. Philadelphia: Saunders Elsevier; 2007. p. 731-3.
- [Result] Jin L, Jin H, Zhang G, Xu G. Changes in coagulation and tissue plasminogen activator after the treatment of cerebral infarction with lumbrokinase. Clin Hemorheol Microcirc. 2000;23(2-4):213-8. PMID 11321442
- [Result] Rey I. Pengaruh pemberian lumbrokinase selama 7 hari terhadap status hiperkoagulasi pada penderita ulkus kaki diabetik. Tugas Akhir Dalam Rangka menyelesaikan Pendidikan Dokter Spesialis Ilmu Penyakit Dalam. FK-USU, Medan. 2009.
- [Result] Trisina J, Sunardi F, Suhartono MT, Tjandrawinata RR. DLBS1033, a protein extract from Lumbricus rubellus, possesses antithrombotic and thrombolytic activities. J Biomed Biotechnol. 2011;2011:519652. doi: 10.1155/2011/519652. Epub 2011 Mar 3. PMID 21403877